CLINICAL TRIAL: NCT03572023
Title: Relationships of Cardiac Structure and Function With Clinical Manifestation of Acute Coronary Syndrome in Patients With Non-obstructed Coronary Arteries
Brief Title: Cardiac Structure, Function, and Clinical Manifestations in MINOCA
Acronym: MINOCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MINOCA
Record Dates: First submitted 2018-06-03; First posted 2018-06-28 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-04

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: Acute coronary syndrome; Non-obstructive coronary artery atherosclerosis; MINOCA; Myocardial infarction; Proinflammatory interleukins; Thrombophilia; Genetic testing; SPECT; MSCT; MRI
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; MINOCA; Thrombophilia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINOCA (Active Comparator): This group will include patients with myocardial infarction with non-obstructive coronary arteries (MINOCA).
  Integrative characterization of MINOCA patients:
  The following interventions will be administered: MSCT, CMR, SPECT, Blood tests, Genetic tests.
  Interventions: Other: Integrative characterization of MINOCA patients
- MI with coronary obstruction (Active Comparator): This group will include patients with myocardial infarction and obstructive coronary arteries.
  Characterization of MI patients with coronary obstruction:
  The following interventions will be administered: MSCT, CMR, SPECT, Blood tests, Genetic tests.
  Interventions: Other: Characterization of MI patients with coronary obstruction

INTERVENTIONS:
Other: Integrative characterization of MINOCA patients — Characterization of MINOCA patients will be based on integrative evaluation of imaging data, blood levels of proinflammatory and anti-inflammatory cytokines, and genetic testing for thrombophilia risk.
  MSCT: Imaging for the presence and vulnerability of coronary plaque as well as plaque disruption.
  CMR: Imaging for identification of myocardial injury (late gadolinium enhancement and myocardial edema) as well as other concomitant findings.
  SPECT: Single-Photon Emission Computed Tomography enable assessment of myocardial perfusion and viability.
  Blood tests.
  Genetic tests.
  Arms: MINOCA
Other: Characterization of MI patients with coronary obstruction — Characterization of patients with myocardial infarction and obstructive atherosclerosis will be based on integrative evaluation of imaging data, blood levels of proinflammatory and anti-inflammatory cytokines, and genetic testing for thrombophilia risk.
  MSCT: Imaging for the presence and vulnerability of coronary plaque as well as plaque disruption.
  CMR: Imaging for identification of myocardial injury (late gadolinium enhancement and myocardial edema) as well as other concomitant findings.
  SPECT: Single-Photon Emission Computed Tomography enable assessment of myocardial perfusion and viability.
  Blood tests.
  Genetic tests.
  Arms: MI with coronary obstruction

SUMMARY:
The purpose of this study is to improve the differential diagnosis and clinical outcomes of acute coronary syndrome with non-obstructive coronary arteries, to investigate the relationship between the structural and functional state of the heart and the clinical course of the disease.

DETAILED DESCRIPTION:
Up to 14% of patients with acute myocardial infarction do not have obstructive changes in the coronary arteries according to invasive coronary angiography (defined as stenosis of > 50% by ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation, 2017). Elevation of highly sensitive Troponin I is a marker of damage to cardiomyocytes, but it is not an underlying mechanism of myocardial damage. Forty patients with acute coronary syndrome are planned to be enrolled in the non-randomized open controlled study. On admission, patients will receive the standard treatment for ACS with and without ST elevation. Within 24 hours, they will undergo diagnostic coronary angiography. In case of nonstenotic atherosclerosis of coronary arteries (normal / stenosis < 50%), patients are planned for cardiac contrast MRI, which will identify both ischemic and non-ischemic causes of acute coronary syndrome; MSCT will be performed to study the coronary arteries and the structure of atherosclerotic plaques; scintigraphy of the myocardium will be performed to characterize the perfusion defect. The frequencies of carrying the genetic alleles associated with the factors that predispose to thrombosis will be studied. Significance of these alleles in the development of thrombosis in acute myocardial infarction will be identified. The profiles of proinflammatory and anti-inflammatory response markers will be determined. Significance of these profiles in the development of acute myocardial infarction in patients with non-obstructive coronary atherosclerosis will be determined in comparison with control group. At one-year follow up, structural and functional characteristics of the heart will be studied again to assess dynamic changes in cardiac state. At one-year follow up, repeated studies will be perform to dynamically assess the structural and functional state of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of enrolment (18 years and older)
* Patients with ACS with and without ST-segment elevation who underwent coronary angiography within 24 h after onset of the disease
* High cardiovascular risk by GRACE Risk Score
* The absence of obstructive coronary atherosclerosis (normal coronary artery / plaques <50%) is based on the results of coronary angiography
* Sinus rhythm on electrocardiogram
* Written informed consent to participate in research

Exclusion Criteria:

* Patients previously undergone endovascular / surgical revascularization of coronary artery
* Severe comorbidity
* Severe renal failure (eGFR < 30)
* Patients with cardiac pacing and claustrophobia
* Contacts / Locations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of unstable plaque occurrence measure | 6 days
  Frequency of occurrence (%) of unstable plaques (including plaque rupture, plaque erosion, and intracoronary thrombus) according to multispiral computed tomography (MSCT) in patients with myocardial infarction with non-obstructive coronary arteries (MINOCA) 6 days after acute coronary syndrome (ACS)

SECONDARY OUTCOMES:
Myocardial perfusion transient defect measure | 1 week
  The magnitude of a transient defect (%) in myocardial perfusion in MINOCA patients in comparison with the control group of patients one week after ACS onset
IL-6 measure | 1 week
  Level of proinflammatory IL-6 in blood plasma in MINOCA patients in comparison with the control group of patients with MI and stenosing arteriosclerosis one week after ACS onset
Pro-thrombophilic allelic variant measure | 3 days
  The frequency of Pro-thrombophilic allelic variant (%), associated with high risk of thrombophilia, in MINOCA patients compared with control group
Frequency of atherosclerosis occurrence measure | 6 days
  Frequency of occurrence (%) of atherosclerosis according to multispiral computed tomography 6 days after acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Ryabov, MD, PhD, Study Director — Tomsk NRMC
Locations (1):
- Vyacheslav Ryabov, Tomsk, Tomsk, Tomskii Region, Russia

IPD SHARING:
Plan to Share IPD: No